CLINICAL TRIAL: NCT07004023
Title: A Randomized, Triple-blind, Placebo Controlled, Cross-over Clinical Trial to Assess the Efficacy of a Single Dose of AlphaWave® L-Theanine on Cognitive Function in Healthy Adults With Moderate Stress
Brief Title: A Clinical Trial to Assess the Efficacy of a Single-dose of AlphaWave® L-Theanine on Cognitive Function in Healthy Adults With Moderate Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ethical Naturals, Inc. (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25ENCCA02
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Function; Moderate Stress
Keywords: Perceived Stress; Moderate Stress; AlphaWave L-Theanine; L-theanine

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind, placebo controlled, cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AlphaWave® L-theanine (Experimental): AlphaWave® L-Theanine, is a dietary supplement containing 200 mg of L-theanine per capsule
  Interventions: Dietary Supplement: AlphaWave® L-Theanine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AlphaWave® L-Theanine — Study staff will provide participants with a single dose of one capsule of AlphaWave® L-Theanine or one placebo capsule with 250 ml of room temperature water.
  Arms: AlphaWave® L-theanine
Other: Placebo — Study staff will provide participants with a single dose of one capsule of AlphaWave® L-Theanine or one placebo capsule with 250 ml of room temperature water.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to to assess the efficacy AlphaWave® L-Theanine on mental acuity/cognitive function and stress relief in healthy adults with moderate stress. The main question it aims to answer is:

Is there a difference in change in mental acuity from pre- to post-dose between AlphaWave® L-Theanine and placebo?

Participants will asked to provided a single dose of one capsule of a single dose of one capsule of AlphaWave® L-Theanine or one placebo capsule with 250 ml of room temperature water, and asked to complete tasks to assess cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 to 60 years of age, inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active during the study
3. Individuals with moderate stress as determined by a score of 14 to 26 on the Perceived Stress Scale
4. Have a regular sleep-wake cycle with a bedtime between 9:00 pm and 12:00 am and receive between 7 and 9 hours of sleep for at least 3 weeks prior to baseline
5. Agrees to avoid caffeine (e.g., tea, coffee, energy drinks) for 12 h prior to post-screening clinic study visits
6. Agrees to avoid alcohol consumption and vigorous physical activity for 24 h prior to post-screening clinic study visits
7. Agrees to avoid first generation anti-allergy medication for 48 h prior to post-screening clinic study visits
8. Willingness to complete assessments and diaries associated with the study and to complete all visits
9. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study
10. Provided voluntary, written, informed consent to participate in the study
11. Healthy as determined by medical history as assessed by the Qualified Investigator (QI)

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, intolerance, or dietary restriction preventing consumption of investigational product or placebo ingredients
3. Self-reported confirmation of any significant neuropsychological condition and/or cognitive impairment (e.g., Schizophrenia, bipolar disorder, post-traumatic stress disorder, brain injury, stroke, neurodegenerative disease, infections, insomnia, depression, epileptic or other seizure-related disorders) that could interfere with study participation as assessed by the QI
4. Self-reported color blindness/weakness as assessed by the QI
5. Current employment that calls for rotating shift work or shift work that will disrupt normal circadian rhythm in the last three weeks as assessed by the QI
6. Unstable metabolic disease or chronic diseases as assessed by the QI
7. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
8. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
9. Type I or Type II diabetes
10. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
11. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
12. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
13. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
14. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
15. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
16. Use of medical cannabinoid products as assessed by the QI
17. Chronic use of cannabinoid products (>2 times/week). Occasional users will be required to washout and abstain for the duration of the study period
18. Regular use of tobacco or nicotine products in the past six months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
19. Alcohol intake average of >2 standard drinks per day as assessed by the QI
20. Alcohol or drug abuse within the last 12 months
21. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (Section 7.3)
22. Participation in other clinical research studies 30 days prior to baseline as assessed by the QI
23. Individuals who are cognitively impaired and/or who are unable to give informed consent
24. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The difference in change in mental acuity from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in mental acuity from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by reaction time using the Computerized Mental Performance Assessment System (COMPASS) tasks.

SECONDARY OUTCOMES:
The difference in change in Cognitive Demand Battery (CDB) from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in Cognitive Demand Battery (CDB) from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by COMPASS.
The difference in change in attention from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in attention from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by COMPASS.
The difference in change in episodic, working and spatial memory from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in episodic, working and spatial memory from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by COMPASS.
The difference in change in psychomotor, processing, and motor speed from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in psychomotor, processing, and motor speed from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by COMPASS.
The difference in change in sustained attention from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in sustained attention speed from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by the Go/No Go assessment.
The difference in change in stress from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in stress from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by the Perceived Stress Scale (PSS). A scale of 1 to 10, with 10 indicating more perceived stress.
The difference in change in stress from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in stress from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by salivary cortisol.
The difference in change in heart rate from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in heart rate from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by salivary cortisol.
The difference in change in blood pressure from pre- to post-dose between AlphaWave® L-Theanine and placebo | 1 hour pre-dose and 1 hour post-dose
  The difference in change in blood pressure from pre- to post-dose between AlphaWave® L-Theanine and placebo as assessed by salivary cortisol.

OTHER OUTCOMES:
Incidence of post-emergent adverse events (AE) | 1 hour pre-dose to 1 hour post-dose
  Incidence of post-emergent adverse events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada